CLINICAL TRIAL: NCT03449212
Title: SOD1 Kinetics Measurements in ALS Patients
Status: Suspended | Type: Observational
Why Stopped: COVID-19 pandemic
Sponsor: Washington University School of Medicine (Other)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Timothy M. Miller, MD, PhD, David Clayson Professor of Neurology, Washington University School of Medicine
Other Study IDs: SOD1-001
Record Dates: First submitted 2018-02-06; First posted 2018-02-28 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Amyotrophic Lateral Sclerosis, Familial; Amyotrophic Lateral Sclerosis, Sporadic
Keywords: SOD1; Amyotrophic Lateral Sclerosis; ALS; Kinetics; Amyotrophic Lateral Sclerosis, Familial; Amyotrophic Lateral Sclerosis, Sporadic
MeSH Terms: conditions — Amyotrophic lateral sclerosis 1; Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, Red Blood Cell (RBC), Cerebral Spinal Fluid (CSF), urine
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- SOD1 ALS
- Sporadic ALS
- Asymptomatic SOD1 gene carriers

SUMMARY:
Washington University in St. Louis is seeking participants with ALS for a study to determine the half-life of the protein SOD1 in the cerebral spinal fluid. Mutations in the SOD1 gene are known to cause some forms of familial ALS. Researchers are developing a treatment to reduce the level of SOD1 in familial ALS, but need to know more about how long SOD1 stays in the body ("half-life") to help determine if the new treatment is effective.

DETAILED DESCRIPTION:
Background: Novel targeted therapeutic strategies are being developed for genetic subsets of ALS, such as those caused by dominantly inherited mutations in the superoxide dismutase 1 gene (SOD1). Investigators have developed an antisense oligonucleotide (ASO) inhibitor of SOD1 biosynthesis for ALS patients who carry mutations in SOD1. This ASO is now ready for clinical trial (ClinicalTrials.gov #NCT02623699). The initial success of the ASO will depend on showing a pharmacodynamics result on SOD1 in participants, and thus a key challenge in applying this targeted therapy involves rigorous examination of pharmacodynamics markers.

The Investigator's previous data suggest that SOD1 in the cerebral spinal fluid (CSF) will be an excellent pharmacodynamics marker for an SOD1-focused therapeutic approach. However, one of the central missing components in understanding SOD1 as a marker is SOD1 CSF half-life data. The half-life of this protein will aid in clinical trial planning since half-life influences the amount of SOD1 protein reduction by ASO and thus dictates the optimal timing of drug administration and CSF collection for pharmacodynamics measures.

Objectives:

* Enroll a total of 86 ALS participants
* Determine the kinetics for total SOD1 protein, as well as the wild type and mutant protein separately
* Determine this in patients with known SOD1 mutation as well as sporadic ALS patients Eligibility
* Adults over age 18
* fALS with confirmed genetic testing showing a mutation in the SOD1 gene; asymptomatic SOD1 gene carriers and sporadic ALS patients.

Measures: The key outcome of this study is to determine the half-life of the SOD1 protein in symptomatic and asymptomatic ALS patients which will provide critical information to inform future therapeutic studies in ALS. For ALS patients, The Investigators will also perform Slow Vital Capacity testing and the ALSFRS-R at the screening visit and at each lumbar puncture visit.

Measures: Participants will have up to 7 in-person visits over 4 months. The study involves labeling or marking SOD1 with a special type of leucine. Leucine is an essential amino acid that is found in the foods we eat. This method involves an overnight stay for a 16 hour intravenous infusion of labeled leucine along with a collection blood and urine followed by 5 lumbar punctures scheduled over the period of 4 months.

At each subsequent visit, subjects will undergo a blood draw, urine collection, lumbar puncture, a questionnaire (ALS Functional Rating Scale) which measures motor function, and a breathing test to determine Slow Vital Capacity (SVC) measurements.

Analysis: In addition to determining the half-life of the SOD1 protein in ALS patients, the Investigators will also analyze the kinetics of wild type SOD1 protein separately from mutant SOD1 protein to determine differences in half life. The Investigators will also compare CSF Tau half-life between ALS patients and controls as a disease specificity control. The Investigators hope to correlate this data with clinical measures which may reveal other important hypotheses regarding SOD1 kinetic rates and disease manifestations.

ELIGIBILITY:
Inclusion Criteria (with exceptions for each group):

* Males or females of any race aged 18 or older
* Positive for SOD1 mutation (SOD1 ALS only)
* Diagnosed with Definite, Probable or Possible ALS in accordance with El Escorial criteria (ALS and SOD1 Positive ALS only)
* Able to hold position and breathe comfortably for the duration of the LP procedure as determined by the LP physician or Nurse Practitioner
* Subjects must be able to provide informed consent

Exclusion Criteria for all groups:

* Invasive ventilator dependence, such as tracheostomy
* Medically unable to undergo lumbar puncture (LP) as determined by the investigator (i.e.,bleeding disorder, allergy to local anesthetics, a skin infection at or near the LP site, or evidence of high intracranial pressure).
* Any active dermatologic disease.
* Any connective tissue disease including systemic lupus erythematous, Sjögren's syndrome, scleroderma or mixed connective tissue disease.
* Any known or suspected abnormal CSF pressure or intracranial/intraspinal tumors.
* Use of anticoagulant medication (eg. warfarin, dalteparin, enoxaparin, rivaroxaban, fondaparinux, dabigatran) that cannot be safely withheld until coagulation parameters have normalized prior to lumbar puncture and for up to a week following the lumbar puncture.
* Blood dyscrasia, abnormal bleeding diathesis, or the use of dialysis for renal failure.
* Clinical judgment of the Site Investigator that the subject would be unable to undergo multiple lumbar punctures.
* Safety lab values greater than 2X the upper limit of normal
* Allergy to Lidocaine
* Pregnancy
* Any contraindication for lumbar puncture

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Known SOD1 positive ALS status, sporadic ALS and SOD1 positive carriers (non-ALS).
Sampling Method: Non-Probability Sample
Enrollment: 86 (Estimated)
Dates: Start 2012-12 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The primary outcome measurement will be the determination of the SOD1 half-life in the CSF of each subject. | Assessed over 121 days
  The half-life of total SOD1 protein will be determined in ALS patients using peptides that do not contain SOD1 mutation. The Investigators will analyze the kinetics of wild type SOD1 protein separately from mutant SOD1 protein using the mutation-containing peptide in order to determine differences in half-life using the stable isotope labeling kinetics (SILK) method of mass spectrometry.

SECONDARY OUTCOMES:
ALS Functional Rating Scale-Revised (ALSFRS-R) | Baseline and weeks 1,2, 4, 9 and 17
  12 questions about patient's ability to function in certain activities of daily living. Each question is out of 4 with 4 being normal and 0 being completely impaired.
Slow Vital Capacity (SVC) | Baseline and weeks 1,2, 4, 9 and 17
  Measurement of the maximum amount of air that can be exhaled following a deep breath.

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University in St. Louis, St Louis, Missouri, United States

REFERENCES:
- [Result] Ly CV, Ireland MD, Self WK, Bollinger J, Jockel-Balsarotti J, Herzog H, Allred P, Miller L, Doyle M, Anez-Bruzual I, Trikamji B, Hyman T, Kung T, Nicholson K, Bucelli RC, Patterson BW, Bateman RJ, Miller TM. Protein kinetics of superoxide dismutase-1 in familial and sporadic amyotrophic lateral sclerosis. Ann Clin Transl Neurol. 2023 Jun;10(6):1012-1024. doi: 10.1002/acn3.51784. Epub 2023 Apr 29. PMID 37119480